CLINICAL TRIAL: NCT03254667
Title: Prospective, Observational Study Brodalumab Compared With Other Therapies in the Treatment of Adults With Moderate-to-Severe Psoriasis Who Are Candidates for Systemic Therapy or Phototherapy in the Course of Actual Clinical Care
Brief Title: LTS of Siliq vs. Other Therapies Treating of Adults With Moderate-to-Severe Psoriasis
Status: Enrolling by invitation | Type: Observational
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: V01-BROA-402
Record Dates: First submitted 2017-08-15; First posted 2017-08-18 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: None Retained — Neutrophil count
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Brodalumad exposed: 1500 subjects exposes to brodalumab
  Interventions: Biological: Brodalumab
- Comparator Subjects: 2000 comparator subjects
  Interventions: Drug: Comparator Drug (non-biologic IL-17 inhibitors)

INTERVENTIONS:
Biological: Brodalumab — Brodalumab
  Groups: Brodalumad exposed
Drug: Comparator Drug (non-biologic IL-17 inhibitors) — Comparator subjects treated with non-biologic IL-17 inhibitors
  Groups: Comparator Subjects

SUMMARY:
Prospective, Observational Study to Assess the Long-Term Safety of Brodalumab Compared with Other Therapies in the Treatment of Adults with Moderate-to-Severe Psoriasis

DETAILED DESCRIPTION:
Prospective, Observational Study to Assess the Long-Term Safety of Brodalumab Compared with Other Therapies in the Treatment of Adults with Moderate-to-Severe Psoriasis Who Are Candidates for Systemic Therapy or Phototherapy in the Course of Actual Clinical Care

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis and main criteria for inclusion: a subject must have moderate to severe psoriasis diagnosed by a dermatologist
2. Must be at least 18 years of age or older
3. Started on or switched to a systemic psoriasis treatment within the previous 12 months. FDA-approved biologic treatments and select non-biologic treatments (eg, methotrexate, cyclosporine, or apremilast only) are permitted.

Exclusion Criteria:

1. The subject is unable or unwilling to provide informed consent to participate in the registry.
2. The subject is participating or planning to participate in a clinical trial with a non-marketed or marketed investigational drug (i.e. Phase I-IV drug trial).
3. The subject is restarting the eligible medication less than 12 months since receiving the last dose.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population consisting of 1500 subjects treated with Brodalumab, and 2000 comparator subjects being treated with a non-biologic IL-17 inhibitor drug.
Sampling Method: Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2030-11-10 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Assess the incidence of malignancy | 8 years
  Assess the incidence of malignancy, excluding non-melanoma skin cancer (NMSC), in adult psoriasis subjects exposed to brodalumab in the course of actual clinical care compared to non-IL-17-inhibitor biologic medications used to treat psoriasis.

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Bhatt, Study Director — Bausch Health
Locations (1):
- Registry, Bridgewater, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided